CLINICAL TRIAL: NCT04081454
Title: The Comfort Ability Workshop: Improving Pain Treatment for Children and Their Families
Brief Title: Comfortability Workshop
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201907083
Record Dates: First submitted 2019-08-17; First posted 2019-09-09 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Educational Status

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with chronic pain
  Interventions: Behavioral: Workshop; Behavioral: Education
- Caregivers of children with chronic pain
  Interventions: Behavioral: Workshop; Behavioral: Education

INTERVENTIONS:
Behavioral: Workshop — one-day (6 hour) program to help children and their parents or caregivers learn how to better manage chronic pain
Behavioral: Education — The parent program includes psychoeducation regarding pain in the context of adolescent development, didactic and vignette-based practice of an adaptive parent communication response style (i.e., reflective listening), and concrete tools for setting up behavior plans to scaffold an adolescent's return to function for school, sleep, daily activities, and exercise. All parents are provided with a take-home workbook inclusive of neuroscience and psychoeducational materials as well as a list of resources to further solidify the information they learned.

SUMMARY:
The Comfort Ability is a fun and interactive one-day (6 hour) program to help children and their parents or caregivers learn how to better manage chronic pain. The program introduces cognitive-behavioral and bio-behavioral pain management strategies to emphasize the mind-body connection and offers non-invasive and non-pharmaceutical strategies for improved pain management. Youth ages 11-18 with chronic or recurrent pain are eligible to sign up for Comfort Ability.

DETAILED DESCRIPTION:
This 1-day, manualized clinical intervention includes a parent group and an adolescent group that run simultaneously, but separately. This program will be offered 4 times per calendar year. The program is 6-hours long and was run at an urban, Midwest children's hospital on a weekend day to maximize accessibility for families. Each group will include between 8 and 12 adolescents (ages 11-17 years) and 15-21 parents. The groups will be staffed by two PhD-level psychologists (one for the parent and one for the adolescent group), a psychology postdoctoral fellow, and nurse practitioner, one or two trained study assistants (e.g., psychology interns, nurse coordinator) who provide support, but not intervention content.

The adolescent program includes motivational interviewing, psychoeducation, and structured activities that emphasize the link between pain, negative cognitions (i.e., catastrophizing), avoidance behaviors, and mood. About one third of the day is devoted to in vivo practice of relaxation-based skills including diaphragmatic breathing, guided imagery, pain-reduction visualization, and biofeedback. Additionally, adolescents participate in several hands-on activities designed to enhance mind-body regulation including mindfulness practice (eating mindfully), art therapy, and aromatherapy. Adolescents complete interactive workbooks throughout the program; at the end of the day, each adolescent works one-on-one with staff to create a written and personalized pain management plan emphasizing the adaptive coping strategies each adolescent preferred during the day. Adolescents were additionally provided with a pain management tool kit inclusive of recorded relaxation exercises, a biofeedback card, and other small tools to enhance their pain management regimen.

The parent program includes psychoeducation regarding pain in the context of adolescent development, didactic and vignette-based practice of an adaptive parent communication response style (i.e., reflective listening), and concrete tools for setting up behavior plans to scaffold an adolescent's return to function for school, sleep, daily activities, and exercise. All parents are provided with a take-home workbook inclusive of neuroscience and psychoeducational materials as well as a list of resources to further solidify the information they learned.

In addition there will be peer support for parents and adolescents in this program. During the 1 day intervention families and youth will be encouraged to share discussions regarding their health journeys. A guest speaker will be invited to both groups sharing their experiences and journey of utilizing psychologically based interventions to assist with reducing pain and stress and associated disability. These speakers have not received training for this portion.

ELIGIBILITY:
Inclusion Criteria:

1. 11 years to 17 years
2. Ability to provide informed consent

Exclusion Criteria:

1. Cognitive Delay that may impact completion of questionnaires and involvement of youth group at workshop.
2. Families without access to internet to complete 1 week, 1 month and 3 month follow up questionnaires.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 11 - 17 with chronic pain and their parents or caregivers
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of this program in change of pain interference: PROMIS | up to 3 months after workshop
  Pediatric pain interference over the past 7 days on scale of 1 - 5. 1=Never, 2=Almost Never, 3=Sometimes, 4=Often, 5=Almost Always
Assess the efficacy of this program in change of pain interference: Pain Self Efficacy Scal - Adolescent | up to 3 months after workshop
  Questionnaire to assess confidence with doing daily tasks when in pain. Scale of 1-5. 1=very sure, 2=pretty sure, 3=in the middle, 4=pretty unsure, 5=very unsure
Assess the efficacy of this program in change of pain interference: Functional Disability Inventory | up to 3 months after workshop
  Questionnaire relating to difficulty of doing regular activities. Scale of 0 - 4. 0=no trouble, 1=a little trouble, 2=some trouble, 3=a lot of trouble, 4=impossible
Assess the efficacy of this program in change of pain interference: Post-Workshop Questionnaire for Parent/Caregiver | up to 3 months after workshop
  Use of questionnaire to measure child's opinion of eductional material during workshop. Scale of 1 -5. 1=Strongly disagree, 2=disagree, 3=unsure, 4=Agree, 5=Strongly Agree
Assess the efficacy of this program in change of pain interference: Pain Catastrophizing Scale | up to 3 months after workshop
  Assess thoughts and feelings when participant is in pain. Scale 0-4. 0=Not at all, 1=to a slight degree, 2=to a moderate degree, 3=to a great degree, 4=all the time
Assess the efficacy of this program in change of pain interference: Pediatric Pain Screen Tool | up to 3 months after workshop
  Assess child's pain location and interference in daily life. Yes/No answers
Assess the efficacy of this program in change of pain interference: Treatment History Questionnaire | up to 2 weeks before workshop
  Questionnaire to capture demographics, medical history, goals of treatment
Assess the efficacy of this program in change of pain interference: Adult Responses to Children's Symptoms | up to 3 months after workshop
  Parent/Caregiver questionnaire to assess child's symptoms. Scale of 0 - 5, with 0=never and 5=often
Assess the efficacy of this program in change of pain interference: Pain Self Efficacy Scale - Child | up to 3 months after workshop
  Questionnaire to assess confidence with doing daily tasks when in pain. Scale of 1-5. 1=very sure, 2=pretty sure, 3=in the middle, 4=pretty unsure, 5=very unsure
Determine if the workshop increases children's pain self-efficacy and improves patients function at our institution: PROMIS | Up to 3 months following workshop
  Pediatric pain interference over the past 7 days on scale of 1 - 5. 1=Never, 2=Almost Never, 3=Sometimes, 4=Often, 5=Almost Always
Determine if the workshop increases children's pain self-efficacy and improves patients function at our institution: Post-Workshop Questionnaire for Parent/Caregiver | up to 3 months after workshop
  Use of questionnaire to measure parent/caregiver's opinion of eductional material during workshop. Scale of 1 -5. 1=Strongly disagree, 2=disagree, 3=unsure, 4=Agree, 5=Strongly Agree
Determine if the workshop increases children's pain self-efficacy and improves patients function at our institution: Functional Disability | Up to 3 months following workshop
  Questionnaire relating to difficulty of doing regular activities. Scale of 0 - 4. 0=no trouble, 1=a little trouble, 2=some trouble, 3=a lot of trouble, 4=impossible
Determine if the workshop increases parental management strategies of their child's pain at our institution: PROMIS | Up to 3 months following workshop
  Pediatric pain interference over the past 7 days on scale of 1 - 5. 1=Never, 2=Almost Never, 3=Sometimes, 4=Often, 5=Almost Always
Determine if the workshop increases parental management strategies of their child's pain at our institution: Pain Evaluation Questionnaire | Up to 3 months following workshop
  Use of questionnaires to measure parental management strategies.
Determine if the workshop increases parental management strategies of their child's pain at our institution: Functional Disability | Up to 3 months following workshop
  Questionnaire relating to difficulty of doing regular activities. Scale of 0 - 4. 0=no trouble, 1=a little trouble, 2=some trouble, 3=a lot of trouble, 4=impossible

CONTACTS AND LOCATIONS:
Overall Officials: Jacob AuBuchon, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coakley R, Wihak T, Kossowsky J, Iversen C, Donado C. The Comfort Ability Pain Management Workshop: A Preliminary, Nonrandomized Investigation of a Brief, Cognitive, Biobehavioral, and Parent Training Intervention for Pediatric Chronic Pain. J Pediatr Psychol. 2018 Apr 1;43(3):252-265. doi: 10.1093/jpepsy/jsx112. PMID 29048506
- [Background] Perquin CW, Hazebroek-Kampschreur AA, Hunfeld JA, van Suijlekom-Smit LW, Passchier J, van der Wouden JC. Chronic pain among children and adolescents: physician consultation and medication use. Clin J Pain. 2000 Sep;16(3):229-35. doi: 10.1097/00002508-200009000-00008. PMID 11014396
- [Background] Roth-Isigkeit A, Thyen U, Raspe HH, Stoven H, Schmucker P. Reports of pain among German children and adolescents: an epidemiological study. Acta Paediatr. 2004 Feb;93(2):258-63. PMID 15046285